CLINICAL TRIAL: NCT05959980
Title: Posterior Cervical Fixation Versus Long-term Cervical Collar for Management of Hirayama Disease: Prospective Randomized Open Blinded Endpoint (PROBE), Phase III Study
Brief Title: Cervical Fixation Surgery Cervical Collar for Management of Hirayama Disease: A Randomized Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Deepti Vibha, Professor, Neurology, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AC-60
Record Dates: First submitted 2023-07-18; First posted 2023-07-25 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Hirayama Disease
Keywords: Hirayama disease; cervical collar; posterior cervical fixation surgery
MeSH Terms: conditions — Amyotrophy, monomelic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical arm (Experimental): Will undergo posterior cervical fixation surgery within 4 weeks of randomization
  Interventions: Procedure: Posterior cervical fixation surgery
- Cervical collar arm (No Intervention): Will be given cervical collar for regular use

INTERVENTIONS:
Procedure: Posterior cervical fixation surgery — These patients will undergo posterior cervical fixation in the form of cervical lateral mass screw fixation in extension without decompression under general anesthesia.
  Arms: Surgical arm

SUMMARY:
The goal of this clinical trial] is to compare cervical collar versus neck stabilization surgery in diagnosed patients of Hirayama disease who have been reporting worsening of problems in the past six months. The main question[s] it aims to answer are:

• Is cervical stabilization surgery (Posterior cervical fixation) superior to conservative management in the form of cervical collar placement in patients with progressive Hirayama disease, observed at six months after intervention

Participants will have equal chance to:

* Undergo cervical fixation surgery
* Cervical collar management The investigators will study and compare the efficacy of both treatments upto six months after intervention

DETAILED DESCRIPTION:
1. Study design:

   Prospective randomized open blinded endpoint (PROBE), phase III study
2. Inclusion criteria:

All the following:

1. Age ≥ 18 years
2. Patients with Hirayama disease as per the following criteria (All of the following) (16):

   1. Clinical evidence of wasting and weakness confined to one limb (EMG evidence of denervation in the opposite limb will not be a reason for exclusion)
   2. Progressive course, or initial progression followed by stationary course; and
   3. No evidence of a compressive lesion of the spinal cord.
3. Disease duration of ≤4 years
4. Progression of clinical symptoms in the past six-months c. Exclusion criteria:

Any of the following:

1) Refusal to consent for randomization 2) Not willing to come for three- and six-months follow-up e. Procedures at baseline:

1. Clinical, electrophysiology and autonomic function assessments:

   After the clinical diagnosis by inclusion criteria, the patients will undergo a detailed clinical examination (as per the case record form (CRF), which includes power, autonomic features, grip strength), and the objective assessment of the electrophysiological parameters
2. Radiological assessment:

   All patients will undergo MR imaging on a 1.5 T MR scanner (Optima 450w, General Electric, Milwaukee, USA), using an 8-channel cervical-thoracic-lumbar array spine coil. The imaging will include axial and sagittal T2-WIs and post-gadolinium T1+C in flexion, neutral and extension positions. In addition, DTI protocol will include sagittal and axial acquisition of cervical cord in neutral position. MR-DTI data will process on a dedicated workstation (Advantage Windows workstation, GE Healthcare, WI, USA) using commercially available software (Functool 14.3.01, GE HealthCare, WI, USA). After co-registration of raw images to correct the motion and distortion artefacts, the ADC and FA images will be generated. The mean, minimum and maximum values of FA and ADC will be recorded from region of maximum cord compression/ T2-hyperintensity.

   The investogators will get a cervical spine radiograph at the time of discharge and at 6 months.
3. Surgical procedure:

The patients who are randomized to undergo posterior cervical fixation will be admitted in Neurosciences Centre, All India Institute of Medical Sciences, New Delhi. These patients will undergo routine preoperative work up, including routine blood investigations and a detailed preanesthetic checkup (PAC). These patients will undergo posterior cervical fixation in the form of cervical lateral mass screw fixation in extension without decompression under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* All the following:

  1. Age ≥ 18 years
  2. Patients with Hirayama disease as per the following criteria (All of the following) (16):

     1. Clinical evidence of wasting and weakness confined to one limb (EMG evidence of denervation in the opposite limb will not be a reason for exclusion)
     2. Progressive course, or initial progression followed by stationary course; and
     3. No evidence of a compressive lesion of the spinal cord.
  3. Disease duration of ≤4 years
  4. Progression of clinical symptoms in the past six-months

Exclusion Criteria:

* Any of the following:

  1. Refusal to consent for randomization
  2. Not willing to come for three- and six-months follow-up

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Odom's criteria score at six months | Six months after intervention

SECONDARY OUTCOMES:
Odom's criteria score at three months | Three months after intervention
interval change in DTI metrics of fractional anisotropy (FA) and apparent diffusion coefficient (ADC) of cervical cord | at six-months post-intervention
Electrophysiological and grip strength | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Deepti Vibha, Principal Investigator — AIIMS, New Delhi
Locations (1):
- Deepti Vibha, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized patient data may be shared on pertinent request